CLINICAL TRIAL: NCT06842706
Title: Prevalence of Drug-resistant Hiv-1 Strains in Patients Experiencing Virologic Failure.(MULTIVIR2025)
Brief Title: Prevalence of Drug-resistant Hiv-1 Strains in Patients Experiencing Virologic Failure. (MULTIVIR2025)
Acronym: MULTIVIR2025
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0788s MULTIVIR2025
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: HIV Infection
Keywords: HIV; drug resistance; antiretrovirals; multi-drug resistant; virological failure
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this cross-sectional, national and multicenter study, the main objective is to determine the prevalence of multi-drug resistant viruses (i.e., viruses that are resistant or possibly resistant to at least one antiretroviral drug from four different therapeutic classes: NRTI, NNRTI, PI, INSTI) among people with HIV 1 (PWH) experiencing virological failure.

DETAILED DESCRIPTION:
Detailed Description:

This is a cross-sectional, national and multicenter study with retrospective and prospective data collection. The study will be conducted in all French virology laboratories that participated in the last quality control for HIV genotypic resistance testing conducted by the ANRS MIE network (n = 42).

Study population All patients treated with antiretrovirals and experiencing virological failure (defined as two consecutive viral loads, at least two weeks apart, greater than 50 copies/mL) can be included in this study.

The study will run for twelve months, with a planned start in 2025. During six months, virologists will be asked to identify all patients meeting the inclusion criteria until they reach 20 patients (for centers following less than 2000 PLWHA) or 40 patients (for centers following more than 2000 PLWHA). Genotypic resistance testing will be performed for all these patients, as recommended by French guidelines. Genotypic resistance testing will always include the amplification of the reverse transcriptase (RT), protease (PR) and integrase (INT), whereas the amplification of gp120, gp41 and/or capsid will only be performed in patients receiving maraviroc, enfuvirtide or lenacapavir, respectively.

Genotypic resistance testing will be performed in each local laboratory, using Sanger or high-throughput sequencing.

Sample size It is estimated that the proportion of patients with multi-drug resistant viruses is between 1 and 5% in this population. Thus, the aim is to include at least 500 patients, which would allow to determine the proportion of multi-drug resistant viruses with an accuracy of 1 to 2%.

With at least 30 participating centers, an expected number of 800 patients should be included. Given the threshold used to define virological failure (50 copies/mL), it is expected that genotypic resistance testing will not be successful in a number of cases. Assuming that all patients with virological failure have viral loads between 51 and 200 copies/mL, and that the success rate for genotypic resistance testing is 63%, the number of patients for whom we would have genotypic data would be 504.

Data collection The virology laboratories will send the list of eligible patients to the associated clinical centers, according to their usual data transfer procedure, so that clinicians can inform the participants and obtain their informed consent. An information form will also be distributed to participants.

A unique identification code will be assigned to each patient that have agreed to this study. An electronic case report form will be used to collect genotypic, clinical and demographic data.

Data analysis Identification of drug resistance-associated mutations will be performed using two different algorithms: Stanford HIVDB (version 9.7, November 2024) and HIV French Resistance (version 35, April 2024).

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) 18 years of age or older.
* Patient who has given his or her consent to participate in the study.
* Patient on antiretroviral therapy for at least six months, with a plasma viral load (VL) greater than 50 copies/mL on at least two consecutive measurements.

Exclusion Criteria:

* Patients opposed to the use of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of people living with HIV (PLHIV) in virological failure, the proportion of participants with virus resistant or possibly resistant to at least one antiretroviral agent from 4 different therapeutic classes: nucleoside reverse transcriptase inhibitor (NRTI), non-nucleoside reverse trancriptase inhibitor (NNRTI), protease inhibitor (PI) and integrase inhibitor (INSTI).
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Drug resistance-associated mutations are those defined in the current ANRS algorithm (https://hivfrenchresistance.org/hiv-french-resitance-tables-of-rules/) and in the current Stanford algorithm (http://hivdb.stanford.edu) at the time of analysis. | Recruitment period: 6 months ·Participation period per participant: 1 day (no follow-up visit) ·Total research period: 12 months · Provisional start date: April 1, 2025 · Provisional end da
  Genotypic resistance to an antiretroviral drug will be interpreted using these two algorithms. Resistance to a therapeutic class will be defined as a resistance, or possible resistance, to all drugs in the class.

CONTACTS AND LOCATIONS:
Overall Officials: Quentin Le Hingrat, DR, Principal Investigator — Bichat-Claude Bernard University Hospital, Paris, AP-HP.Nord; Constance Delaugerre, PR, Principal Investigator — Service de Virologie Hôpital Saint-Louis, AP-HP.Nord 1 avenue Claude Vellefaux, 75010 Paris

IPD SHARING:
Plan to Share IPD: No